CLINICAL TRIAL: NCT04543318
Title: Using the Deep Temporal Nerves Versus the Masseteric Nerve for Correction of Eyelid Paresis Caused by Facial Nerve Affection. A Comparative Clinical Study.
Brief Title: Using the Deep Temporal Nerves Versus the Masseteric Nerve for Correction of Eyelid Paresis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Refaat Ahmed Abdelkarim, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCT04543318
Record Dates: First submitted 2020-09-03; First posted 2020-09-10 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Facial Paresis
MeSH Terms: conditions — Facial Paralysis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep temporal nerves group (Experimental): this group will use deep temporal nerves for reactivation of affected upper facial nerve branch
  Interventions: Procedure: Deep temporal nerves
- Masseteric nerve group (Active Comparator): this group will use masseteric nerve for reactivation of affected upper facial nerve branch (gold standard)
  Interventions: Procedure: massteric nerve

INTERVENTIONS:
Procedure: Deep temporal nerves — Surgical procedure:
  Group A Exploration on the affected side a facelift-type incision will be performed, and an anterior subcutaneous flap is then will be lifted for several centimetres. In the inferior zygomatic region, the plane of elevation is deepened into the sub-SMAS plane and a composite flap elevated for several centimetres. Following elevation in this plane, the distal facial nerve branches will be identified. The distal portion of the zygomatic nerve is usually located midway between the oral commissure and the helical root. and was confirmed by nerve stimulator.
  The deep temporal fascia and temporalis muscle will be incised along the temporal fusion line and will be reflected from the skull to expose the divisions of the deep temporal nerves and the longest branch was traced and prepared for anastomosis end to end with the zygomatic branch after confirming the eyelid supply.
  Arms: Deep temporal nerves group
Procedure: massteric nerve — group B The same procedure as group A except tracing the masseteric nerve related to masseter muscle and anastomosis will be the same
  Arms: Masseteric nerve group

SUMMARY:
The return of eyelid function and facial expression in Patients with facial nerve affection is very important for quality of life. Eyelid dysfunction leads to drying and ulceration of cornea which may lead to permanent vision loss.

Facial paralysis is distinguished into two main groups according to the presence or absence of facial fibrillations at needle Electromyography. Recent paralysis, mainly lasting less than two years generally show these signs and are eligible for reactivation of facial nerve by anastomosing it to a donor one (early facial reanimation).

The masseteric nerve (motor branch of trigeminal nerve ) is a reliable donor nerve on early facial reanimation.

The deep temporal nerves are motor branches of trigeminal nerve which have some advantage over masseteric nerve as they are longer and reach the zygomatic and frontal branch of facial nerve and it can reach the eyelid and eyebrow to be used for direct neurotization and it supplies temporalis muscle which is an expandable muscle with little effect on mastication and it was reported that they can restore blinking.

So on this study we examine the advantages and disadvantages of both nerves to develop a protocol for use of both especially on eyelid reanimation and restoration of blinking on upper facial segment paresis

DETAILED DESCRIPTION:
Type of the study: Prospective Interventional Study (clinical trial)

Intervention Model Description:

Patients will be randomized into two groups according to the surgical procedure performed as follows:

* Group A: Deep temporal nerves.
* Group B: Masseteric nerve.

Allocation and Randomization:

Twenty-four patients will be randomly assigned to Group A or Group B (2 equal groups).

Simple randomization will be performed before surgery by a research nurse using the closed-envelope technique.

Twenty-four closed envelopes will be used, each 12 of them carries one of the 2 groups. Closed envelope will be randomly withdrawn the night before surgery to assign the patient to his specific group.

Study Setting: Plastic and Reconstructive Surgery Department, Assuit University Hospital

Study subjects:

Inclusion criteria:

1. Facial nerve paresis with upper eyelid affection.
2. Patients are generally fit with no other disease interfere with microsurgery.
3. Electromyography of eyelid showing fibrillations. b. Exclusion criteria:

1. Patient with other medical or mental disease causing generalized paralysis. 2. Syndromic cases. 3. Patients are generally unfit or with any disease interfere with microsurgery.

4. Electromyography of eyelid showing no fibrillations.

Sample Size Calculation: 24 Sample size was calculated using G power program version 3.1.9.4 (6) in order to detect a significant difference in mean of palpebral fissure height (one of main assessed outcomes in the study ) between two groups under the study , assumed effect size 0.6 based on clinical assumption ( novel study ), α error 0.3 , power 0.80, and allocation ratio 1: 1.

Twenty-two patient plus 10% for dropouts to make total twenty-four (12 patient for every group).

Study tools

All patients in this study are subjected to:

Pre-operative Assessment:

1. Patient history.
2. All patients will do preoperative clinical and neurophysiological assessments of mimetic muscle function and donor nerve status (the ipsilateral deep temporal nerve. The neurophysiological tests will include needle Electromyography (EMG) for recruitment of residual motor unit action potential. If there are no fibrillations patients will have another surgical procedure.
3. The trigeminal motor component will be tested by palpating the temporalis muscle during chewing and via needle EMG of the temporalis muscle to verify availability as a donor motor nerve.
4. Photographic documentation preoperative using standardized frontal face view and adding a scale to photo to measure the palpebral fissure size during three states normal eye opening, resting eye closure and forced eye closure using ImageJ (image processing and analysis in java) computer software (7).
5. Ophthalmological assessment of the affected eye for detection of redness, ulcer, etc.

Surgical procedure:

Group A We will avoid the use of muscle relaxants to induce anaesthesia and employ an electro-stimulator to identify the deep temporal nerves and the facial nerve branches supplying the eyelid on the affected side.

Exploration on the affected side a facelift-type incision will be performed, and an anterior subcutaneous flap is then will be lifted for several centimetres. In the inferior zygomatic region, the plane of elevation is deepened into the sub-SMAS plane and a composite flap elevated for several centimetres. Following elevation in this plane, the distal facial nerve branches will be identified. The distal portion of the zygomatic nerve is usually located midway between the oral commissure and the helical root. and was confirmed by nerve stimulator.

The deep temporal fascia and temporalis muscle will be incised along the temporal fusion line and will be reflected from the skull to expose the divisions of the deep temporal nerves and the longest branch was traced and prepared for anastomosis end to end with the zygomatic branch after confirming the eyelid supply(8).

Then suction drain will be put and will be removed after 24 hours. Group B The same procedure except tracing the masseteric nerve related to masseter muscle and anastomosis will be the same (9).

Post-operative All patient will receive physiotherapy and post-operative follow up to detect any wound complication.

Evaluation (After 6 months from the operation)

1. Photo documentation: measurement of the palpebral fissure size during three states normal eye opening, resting eye closure , forced eye closure will be done adding eye closure during mastication to compare with preoperative resting eye closure measure using ImageJ (image processing and analysis in java) computer software(7).
2. Donor site morbidity.
3. Follow up Ophthalmological assessment.

Complications:

1. General surgical complication.
2. General complication due to general anaesthesia.
3. Specific complication:

   1. Delayed healing of nerve anastomosis.
   2. Affection of mastication.
   3. No postoperative improvement.

Research outcome measures:

a. Primary (main): Comparing the outcomes on palpebral fissure size between the deep temporal group and the masseteric group after 6 months from the surgery.

a. Secondary (subsidiary):

1. Procedure-related morbidity and mortality.
2. Operative time and hospital stay.

ELIGIBILITY:
Inclusion Criteria:

1. Facial nerve paresis with upper eyelid affection.
2. Patients are generally fit with no other disease interfere with microsurgery. 3.Electromyography of eyelid showing fibrillations.

Exclusion Criteria:

1. Patient with other medical or mental disease causing generalized paralysis.
2. Syndromic cases.
3. Patients are generally unfit or with any disease interfere with microsurgery.
4. Electromyography of eyelid showing no fibrillations.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Palpebral fissure size | 6 months after surgery
  Comparing the outcomes on palpebral fissure size between the deep temporal group and the masseteric group after 6 months from the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abdelkarim, MD, Principal Investigator — Faculty of Medicine,Assiut university,Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Okochi M, Ueda K, Okochi H, Asai E, Sakaba T, Kajikawa A. Facial reanimation using hypoglossal-facial neurorrhaphy with end-to-side coaptation between the jump interpositional nerve graft and hypoglossal nerve: Outcome and duration of preoperative paralysis. Microsurgery. 2016 Sep;36(6):460-6. doi: 10.1002/micr.22393. Epub 2015 Aug 28. PMID 26316293
- [Background] Okochi M, Okochi H, Asai E, Sakaba T, Ueda K. Eyelid reanimation using crossface nerve graft: Relationship between surgical outcome and preoperative paralysis duration. Microsurgery. 2018 May;38(4):375-380. doi: 10.1002/micr.30264. Epub 2017 Nov 10. PMID 29125661
- [Background] Terzis JK, Tzafetta K. The "babysitter" procedure: minihypoglossal to facial nerve transfer and cross-facial nerve grafting. Plast Reconstr Surg. 2009 Mar;123(3):865-876. doi: 10.1097/PRS.0b013e31819ba4bb. PMID 19319050
- [Background] Biglioli F, Frigerio A, Colombo V, Colletti G, Rabbiosi D, Mortini P, Dalla Toffola E, Lozza A, Brusati R. Masseteric-facial nerve anastomosis for early facial reanimation. J Craniomaxillofac Surg. 2012 Feb;40(2):149-55. doi: 10.1016/j.jcms.2011.03.005. Epub 2011 Apr 3. PMID 21463951
- [Background] Karagoz H, Ozturk S, Malkoc I, Diyarbakir S, Demirkan F. Anatomy of the Anterior Deep Temporal Nerve: Implications for Neurotization in Blinking Restoration in Facial Paralysis. Ann Plast Surg. 2015 Sep;75(3):316-8. doi: 10.1097/SAP.0000000000000552. PMID 26101977
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Schneider CA, Rasband WS, Eliceiri KW. NIH Image to ImageJ: 25 years of image analysis. Nat Methods. 2012 Jul;9(7):671-5. doi: 10.1038/nmeth.2089. PMID 22930834
- [Background] Dauwe PB, Hembd A, De La Concha-Blankenagel E, Saba S, White C, Cardenas-Mejia A, Rozen SM. The Deep Temporal Nerve Transfer: An Anatomical Feasibility Study and Implications for Upper Facial Reanimation. Plast Reconstr Surg. 2016 Sep;138(3):498e-505e. doi: 10.1097/PRS.0000000000002482. PMID 27556625
- [Background] Gray ML, Hu S, Gorbea E, Mashkevich G. Masseteric-zygomatic nerve transfer for the management of eye closure-smile excursion synkinesis. Am J Otolaryngol. 2020 Jul-Aug;41(4):102479. doi: 10.1016/j.amjoto.2020.102479. Epub 2020 Apr 4. PMID 32359868